CLINICAL TRIAL: NCT03513211
Title: A Phase I/II Study of Hydroxychloroquine and Itraconazole as Therapy for Men With Androgen Normalised Prostate Cancer
Brief Title: Phase I/II Study of Hydroxychloroquine With Itraconazole With Biochemically Recurrent Prostate Cancer
Acronym: HITMAN-PC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St Vincent's Hospital, Sydney (Other)
Responsible Party: Principal Investigator, Anthony Joshua, FRACP, Head of Medical Oncology, The Kinghorn Cancer Centre, St Vincent's Hospital, Sydney
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HITMAN
Record Dates: First submitted 2018-04-17; First posted 2018-05-01 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Prostate Cancer
Keywords: Biochemically recurrent prostate cancer; Hormone sensitive prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Phase I intra-patient dose escalation study Phase II Simon 2-stage cohort expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose escalation arm (Experimental): Suba-itraconazole in combination dose escalating hydroxychloroquine H
  Interventions: Drug: SUBA-itraconazole; Drug: Hydroxychloroquine
- Phase II: Dose expansion arm (Experimental): Suba-itraconazole with recommended phase II dose of hydroxychloroquine as determined by phase I arm.
  Interventions: Drug: SUBA-itraconazole; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: SUBA-itraconazole — 150mg PO BD
Drug: Hydroxychloroquine — Escalating doses in Rolling 6 Phase I

SUMMARY:
Recent pre-clinical work has suggested that Itraconazole has an anti-cancer effect that works synergistically with hydroxychloroquine. This may delay the need for androgen deprivation therapy (ADT) and its associated toxicities in men with biochemically recurrent (BCR) prostate cancer. This study aims to determine feasibility, safety and efficacy of suba-itraconazole (SI) in combination with hydroxychloroquine (HQ) in the treatment of biochemically recurrent (BCR) prostate cancer as means of delaying time to commencement of androgen deprivation therapy.

DETAILED DESCRIPTION:
A rising PSA following treatment with definitive prostatectomy or radiation therapy for localised prostate cancer represents biochemical relapse (BCR), a disease state for which there is no consensus on optimal management. A proportion of men with BCR will go on to develop metastatic disease but there may be a prolonged period of time between biochemical recurrence and overt clinic progression. Though androgen deprivation therapy (ADT) may prolong metastasis-free survival, it comes at a cost of significant morbidity. Thus substantial efforts are underway to find treatments that may delay the need for ADT while maintaining quality of life in men with BCR prostate cancer.

Autophagy inhibitors given in combination with cytotoxic agents have been found to suppress tumour growth and trigger cell death to a greater extent than chemotherapy alone, both in vitro and in vivo. Such inhibitors include the anti-malarial drug chloroquine (CQ) and its derivative, hydroxychloroquine (HCQ). Taken together, autophagy may represent a major mechanism for treatment resistance and thus, represents a potential novel therapeutic target. Moreover, hydroxychloroquine has shown modest activity as a single agent in men with BCR prostate cancer.

The antifungal drug itraconazole has shown some activity in prostate cancer. These effects are attributed to inhibitory effects on endothelial cell proliferation and angiogenesis, mTOR inhibition through effects on intracellular cholesterol trafficking, hedgehog pathway inhibition and induction of autophagy. With regards to cholesterol trafficking, itraconazole causes depletion of plasma membrane cholesterol and cholesterol trapping in the late endosomes and lysosomes in part through inhibition of the cholesterol transporter NPC1.

Pre-clinical studies have shown enhanced death of prostate cancer cells with treatment of itraconazole combined with hydroxychloroquine. This treatment causes a dramatic increase in the accumulation of free cholesterol with a phenotype reminiscent of Niemann-Pick Syndrome, a neurodegenerative disease characterised by accumulation of free cholesterol in late endosomes/lysosomes due to mutations in NPC1 and NPC2. The investigators hypothesise that itraconazole synergises with hydroxychloroquine to induce sequestration of cholesterol in the lysosomes while inhibiting autophagy thereby inducing cell death through oxidation of the excess cholesterol and cell dysfunction as a result of the inaccessibility of the cholesterol. This mechanism may be particularly potent in androgen sensitive prostate cancer where cholesterol use is destined for androgen synthesis.

Non-castrating treatments for BCR and metastatic prostate cancer are an area of unmet need. The aim of this study is to assess the tolerability, safety and efficacy of hydroxychloroquine in combination with itraconazole as a strategy to delay time to ADT commencement in men with BCR prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Males ≥ 18 years of age with histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features
2. Prostate cancer initially treated by radical prostatectomy, radiotherapy (including brachytherapy) or both, with curative intent
3. PSA ≥ 1 ng/ml with at least two sequential rises at least 1 week apart according to PCWG3.
4. Serum testosterone ≥ 5 nmol/L
5. QTc ≤ 470 msec using Fridericia correction formula
6. Adequate bone marrow function with platelets ≥ 100 x 10^9/L, ANC ≥ 1.5 x 10^9/L, Hb ≥ 100 g/L in the absence of transfusion
7. Adequate liver function with ALT/AST < 1.5 x ULN, bilirubin < 1.5 x ULN
8. Adequate renal function with creatinine clearance > 50 ml/min
9. ECOG Performance Status ≤ 1
10. Able to start study treatment within 28 days of consent
11. Willing and able to comply with all study requirements, including treatment (e.g. able to swallow tablets), timing and/or nature of required assessments
12. Signed, written informed consent

Exclusion Criteria:

1. Contraindications to investigational product including hypersensitivity, treatment with any CYP3A4 inducer or inhibitor or known G6PD deficiency. If on a statin, must be changed to rosuvastatin or ceased, as appropriate
2. Evidence of metastatic disease on conventional WBBS or CT. However low volume regional nodes (≤ N1, up to the aortic bifurcation) may be accepted in asymptomatic patients.
3. PSA doubling time ≤ 3 months calculated using MSKCC calculator (https://www.mskcc.org/nomograms//prostate/psa-doubling-time)
4. Prior systemic therapy for advanced cancer prostate cancer such as hormonal therapy or chemotherapy; neo/adjuvant hormonal therapy allowed if ≤ 24 months total duration and ceased ≥ 12 months prior to enrolment
5. Life expectancy of ≤ 1 year
6. History of another invasive cancer within 3 years before screening with the exception of fully treated cancer with remote probability of recurrence
7. Concurrent illness, including severe infection that may jeopardize the ability of the patient to undergo the procedures outlined in this protocol with reasonable safety
8. Use of hydroxychloroquine and/or itraconazole for any indication in the preceding 2 years or at any time for treatment of prostate cancer.

8. Serious medical or psychiatric conditions that might limit the ability of the patient to comply with the protocol.

9. Men must have been surgically sterilised or use a barrier method of contraception.

10. Pre-existing retinopathy, keratopathy or other ocular pathologies that, in the opinion of an ophthalmologist would put the patient at risk of hydroxychloroquine induced retinopathy 11. History of cardiac failure or recent history if ischaemic heart disease (<2 years)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Determination of Recommended Phase II Dose of Hydroxychloroquine in combination with Suba-itraconazole | 6 months
  Recommended Phase II Dose

SECONDARY OUTCOMES:
PSA response rate | 1 year
  Fall in PSA >/=50% from baseline
Composite safety | 1 year
  Rate of adverse events defined by CTCAE criteria
Time to ADT commencement | 1 year
  Time to start of ADT
Metastasis-free survival | 1 year
  Time from commencement of treatment to first metastatic lesion on CT or WBBS

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Joshua, MBBS(Hons) PhD, Principal Investigator — St Vincent's Hospital, Sydney
Locations (1):
- St Vincent's Hospital, Darlinghurst, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suzman DL, Antonarakis ES. High-dose itraconazole as a noncastrating therapy for a patient with biochemically recurrent prostate cancer. Clin Genitourin Cancer. 2014 Apr;12(2):e51-3. doi: 10.1016/j.clgc.2013.11.015. Epub 2013 Nov 14. No abstract available. PMID 24332506
- [Background] Farrow JM, Yang JC, Evans CP. Autophagy as a modulator and target in prostate cancer. Nat Rev Urol. 2014 Sep;11(9):508-16. doi: 10.1038/nrurol.2014.196. Epub 2014 Aug 19. PMID 25134829